CLINICAL TRIAL: NCT05514275
Title: Radiotherapy Combined With Recombinant Human Endostatin and Capecitabine for Patients With Nasopharyngeal Carcinoma Resistant to Induction Chemotherapy
Brief Title: Radiotherapy Combined With Endostatin and Capecitabine for NPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Jin Ting, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCECNPC
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Radiotherapy; Endostatin; Capecitabine
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Endostatins; Capecitabine

STUDY DESIGN:
Intervention Model Description: Radiotherapy Combined With Endostatin and Capecitabine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endostatin and Capecitabine (Experimental): Patients received radiotherapy Combined With Endostatin and Capecitabine
  Interventions: Drug: Endostatin and Capecitabine

INTERVENTIONS:
Drug: Endostatin and Capecitabine — Patients received radiotherapy Combined With Endostatin(37.5mg/m2, continuous intravenous infusion for 120h, D-7, D8, D22, D36) and Capecitabine( 650 mg/m2 bid, orally, d1-21, every 3 weeks as a cycle for 17 cycles)

SUMMARY:
Radiotherapy combined with recombinant human endostatin and capecitabine for patients with nasopharyngeal carcinoma (NPC) resistant to induction chemotherapy.

DETAILED DESCRIPTION:
This study was a single-arm, open-label, phase II study of radiotherapy combined with recombinant human endostatin and capecitabine for patients with nasopharyngeal carcinoma (NPC) resistant to induction chemotherapy. fourty-one patients of locally advanced NPC resistant to induction chemotherapy were enrolled. Patients received radiotherapy combined with recombinant human endostatin and capecitabine. The primary endpoint was Recurrence free survival (RFS). Secondary goals included overall survival (OS), distant metastasis-free survival (DMFS), Local-regional free survival (LRFS); adverse events (AEs) and severe adverse events (SAE); safety and quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO) histologically type).

Tumor staged as T3-4N1/N2-3 (according to the 8th American Joint Commission on Cancer edition).

No evidence of distant metastasis (M0). Satisfactory performance status: Karnofsky scale (KPS) > 70. Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.

Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.

Adequate renal function: creatinine clearance ≥60 ml/min. Patients must be informed of the investigational nature of this study and give written informed consent.

unsatisfactory tumor response (stable or progressive disease) after neoadjuvant chemotherapy (NACT)

Exclusion Criteria:

WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.

Treatment with palliative intent. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.

Pregnancy or lactation. History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).

Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

satisfactory tumor response (complete response or partial response) after neoadjuvant chemotherapy (NACT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) | 3 years
  calculated from the date of randomisation to the date of locoregional failure, distant failure, or death from any cause, whichever occurred first

SECONDARY OUTCOMES:
overall survival (OS) | 5 years
  calculated from date of randomisation to death
distant metastasis-free survival (DMFS) | 3 years
  calculated from date of randomisation to the first distant failure
Local-regional free survival (LRFS) | 3 years
  calculated from date of randomisation to the first Local-regional failure
adverse events (AEs) and severe adverse events (SAE) | 5 years
  graded according to NCI CTCAE v5.0
quality of life (QoL) | 3 years
  the change of QoL from randomization to 12 months after chemoradiation, graded according to EORTC QLQ-C30 V3.0

CONTACTS AND LOCATIONS:
Overall Officials: Ting Jin, MD, Study Chair — Department of Radiation Oncology, Zhejiang Cancer Hospital
Locations (7):
- China (7):
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - the First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua Central Hospital, Jinhua, Zhejiang
  - The Central Hospital of Lishui City, Lishui, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Ningbo Medical Center Lihuili Eastern Hospital, Ningbo, Zhejiang
  - People's Hospital of Quzhou, Quzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided